CLINICAL TRIAL: NCT02498028
Title: Clinical Outcome After Anterior Cervical Decompression and Fusion and Cervical Total Disc Replacement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Dr. Yorck Rommelspacher, Dr. med. Yorck Rommelspacher, University Hospital, Bonn
Other Study IDs: UKBORTYC01
Record Dates: First submitted 2015-05-02; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Cervical Disc Disorders
Keywords: cervical fusion; cervical arthroplasty; cervicobrachial pain
MeSH Terms: conditions — Klippel-Feil Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cervical Fusion: patients with anterior cerivical decompression and fusion
  Interventions: Procedure: Cervical Fusion
- Cervical Disc Prostheses: patients with cervical total disc replacement
  Interventions: Procedure: Cervical disc Prostheses

INTERVENTIONS:
Procedure: Cervical Fusion — Cervical Fusion is performed with a titanium cage (Company Peter Brehm, Weisendorf, Germany) and a plating system (Company Aesculap, ABC plating system, Tuttlingen, Germany)
  Groups: Cervical Fusion
Procedure: Cervical disc Prostheses — The total disc replacement is performed with eiter a Freedom® Cervical Disc, AxioMed Spine Corporation, Garfield Heights, Ohio, USA or Active® C, Company, Aesculap, Tuttlingen, Germany
  Groups: Cervical Disc Prostheses

SUMMARY:
The aim of this study is to examine the clinical outcome after anterior cervical decompression and fusion, and cervical disc prostheses in general. Additionally these two surgical methods for degenerative diseases of the cercival spine are analyzed comparatively in order to see whether one procedure should be preferred.

DETAILED DESCRIPTION:
The study population consists of patients who are suffering from neck and cervicobrachial pain because of degenerative diseases of the cervical spine. In that population conservative treatment such as analgesia and physiotherapy is no more sufficient, so that surgery is necessary. For surgical treatment are chosen either total disc replacement with an cervical disc prostheses or anterior cervical decompression and fusion.

In the context of this work the clinical success of these surgical methods should be analasied by means of the neck disability index (NDI), the visual analogue scale (VAS) in centimeter, clinical examinations, the satisfaction of patients with the surgery and the occurrence of adverse events. The included patients are examined and seen before and after the surgery.

Furthermore the two different methods are compared to each other in order to detect a possible advantage of one type of surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have to undergo surgery such as spondylodesis or disc prosthesis of the cervical spine because of degenerative diseases and who have been operated in the University Hospital of Bonn between 2011 and 2015.

Exclusion Criteria:

* Patients under the age of 18 years
* Pregnant women
* Patients who are not willing to participate in the study
* Patients unable to take part in the study because of any other known restriction or incompatibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the University Hospital of Bonn who are suffering from neck and cervicobrachial pain that cannot be treated anymore by conservative methods and have to undergo surgery such as cervical fusion or cevical disc arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change in pain as assessed by VAS | Preoperative (baseline day 0), Follow up (24 months)
  Pain objectified by the VAS

SECONDARY OUTCOMES:
Change in Neck disability Index | Preoperative (baseline day 0), Follow up (24 months)
  Restrictions in patients' daily life objecitfied by the NDI (neck disabiliy index)

OTHER OUTCOMES:
Adverse events/ postoperative complications | postoperative until Follow up in 24 months
  Adverse events as for example reoperation because of adjacent segment degeneration or implant loosening
Change in pharmacological pain management, WHO Scale | Preoperative (baseline day 0), Follow up (24 months)
  Pain objectified by the analgesia scheme of the World Health Organisation
Patient satisfaction with the surgical procedure | Follow up (24 months)
  Satisfaction of patients with the result of the operation assessed by grades 1-6

CONTACTS AND LOCATIONS:
Overall Officials: Yorck Rommelspacher, Dr. med, Principal Investigator — University Hospital, Bonn
Locations (2):
- Germany (2):
  - Universitiy Hospital of Bonn, Bonn, North Rhine-Westphalia
  - University hospital Bonn, Bonn